CLINICAL TRIAL: NCT03919500
Title: Erythropoietin Protects Very Preterm Infants Against Necrotizing Enterocolitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhengzhou University (Other)
Collaborators: Zhengzhou Children's Hospital, China (Other); The First Affiliated Hospital of Zhengzhou University (Other); Women and Children Health Care Center of Luoyang, China (Unknown); Göteborg University (Other)
Responsible Party: Principal Investigator, Changlian Zhu, Director, Clinical research center of Third Affiliated Hospitial, Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HN-2014002
Record Dates: First submitted 2019-04-11; First posted 2019-04-18 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Premature Infant
Keywords: Preterm infant; Necrotizing enterocolitis; Erythropoietin; Neurodevelopment
MeSH Terms: conditions — Premature Birth; Enterocolitis, Necrotizing | interventions — epoetin beta; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erythropoietin (Experimental): Infants in the EPO group are given EPO 500IU/kg dissolved in 2 ml saline intravenously every other day for 2 weeks starting within 72 hours after birth.
  Interventions: Drug: EPO
- Normal saline (Placebo Comparator): Infants in the control group are given normal saline intravenously with the same volume as EPO every other day for 2 weeks.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: EPO — Infants in EPO group are administered 500IU/kg intravenously within 72 hours after birth every other day for 2 weeks.
  Other Names: Epoetin Beta
  Arms: Erythropoietin
Drug: Normal saline — Infants in control group are administered normal saline with the same volume and period as EPO.
  Arms: Normal saline

SUMMARY:
This study evaluates the effect of repeated low-dose erythropoietin (EPO) treatment on necrotizing enterocolitis (NEC) in very preterm infants. Half of participants will receive EPO, while the other half will receive a placebo.

DETAILED DESCRIPTION:
NEC is one of the most severe complications in preterm neonates and is associated with high morbility and mortality. Studies have reported that EPO treatment decreases the incidence and severity of experimental NEC in animal models. Evidence from previous clinical studies about the effect of EPO treatment against NEC have all been hampered by small numbers of patients. The study is to investigate whether repeated low-dose EPO protects against NEC. Preterm infants with gestational age ≤32 weeks who are admitted to neonatal intensive care units within 72 hours after birth are randomized to EPO (500IU/kg, intravenously every other day for 2 weeks) or control group (the same volume of saline). Primary outcome is the incidence of NEC at 36 weeks of corrected age. Secondary outcome is growth and neurodevelopment at 18 months of corrected age in infants with NEC.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with gestation age ≤ 32weeks
* Within 72 hours after birth
* Written informed consent obtained from parents

Exclusion Criteria:

* Genetic or metabolic diseases
* Congenital abnormalities
* Polycythemia
* Intracranial hemorrhage grade III/IV
* Unstable vital signs (such as respiration and circulation failure)

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1285 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Incidence of NEC | At 36 weeks of corrected age
  To compare the incidence of NEC between EPO group and control group at 36 weeks of corrected age

SECONDARY OUTCOMES:
Incidence of low height in patients with NEC | At corrected age of 18 months
  To compare the incidence of low height in patients with NEC between EPO and control groups via the Standardized Growth Curve for Chinese Children at 18 months of corrected age.
Incidence of low weight in patients with NEC | At corrected age of 18 months
  To compare the incidence of low weight in patients with NEC between EPO and control group via the Standardized Growth Curve for Chinese Children at 18 months of corrected age.
Incidence of low head circumference in patients with NEC | At corrected age of 18 months
  To compare the incidence of low head circumference in patients with NEC between EPO and control group via the Standardized Growth Curve for Chinese Children at 18 months of corrected age.
Incidence of MDI<70 in patients with NEC | At corrected age of 18 months
  To compare the incidence of MDI<70 in patients with NEC between EPO and control group via Bayley Scales of Infant Development (second edition) at 18 months of corrected age.
Incidence of cerebral palsy in patients with NEC | At corrected age of 18 months
  To compare the incidence of cerebral palsy in patients with NEC between EPO and control group at 18 months of corrected age.
Incidence of blindness in patients with NEC | At corrected age of 18 months
  To compare the incidence of blindness in patients with NEC between EPO and control group via visual acuity at 18 months of corrected age.
Incidence of deafness in patients with NEC | At corrected age of 18 months
  To compare the incidence of deafness in patients with NEC between EPO and control group via auditory brainstem response measurement at 18 months of corrected age.
The effect of EPO treatment on blood messenger RNA (mRNA) expression | At 3 weeks after birth
  To investigate different mRNA expression between EPO and control group, peripheral venous blood of preterm infants after EPO treatment will be collected in both EPO group and control group, and the transcriptome of the premature infant blood will be assayed by RNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Changlian Zhu, PhD, Study Chair — Third Affiliated Hospital of Zhengzhou University
Locations (1):
- Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be assessed by sponsor. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Sun H, Song J, Kang W, Wang Y, Sun X, Zhou C, Xiong H, Xu F, Li M, Zhang X, Yu Z, Peng X, Li B, Xu Y, Xing S, Wang X, Zhu C. Effect of early prophylactic low-dose recombinant human erythropoietin on retinopathy of prematurity in very preterm infants. J Transl Med. 2020 Oct 19;18(1):397. doi: 10.1186/s12967-020-02562-y. PMID 33076939
- [Derived] Wang Y, Song J, Sun H, Xu F, Li K, Nie C, Zhang X, Peng X, Xia L, Shen Z, Yuan X, Zhang S, Ding X, Zhang Y, Kang W, Qian L, Zhou W, Wang X, Cheng X, Zhu C. Erythropoietin prevents necrotizing enterocolitis in very preterm infants: a randomized controlled trial. J Transl Med. 2020 Aug 8;18(1):308. doi: 10.1186/s12967-020-02459-w. PMID 32771013